CLINICAL TRIAL: NCT02772432
Title: Development of a Resiliency Training Program for Parents of Children With Specific Learning Disabilities
Acronym: SPLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Marino Foundation (Unknown)
Responsible Party: Principal Investigator, Elyse Park, PhD, Associate Professor in Psychiatry (HMS), Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016P000423
Record Dates: First submitted 2016-05-12; First posted 2016-05-13 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Stress
Keywords: resiliency training; parenting; special learning disability

STUDY DESIGN:
Intervention Model Description: Patients are assigned to the immediate or wait-list control intervention group.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3RP treatment (Experimental): An adapted version of the Relaxation Response Resiliency Program (3RP) for parents of children with specific learning disabilities. The adapted program incorporates the three prongs of the 3RP: RR elicitation, stress awareness, and adaptive strategies.
  Interventions: Behavioral: Relaxation Response Resiliency Training for Parents of SPLD
- Waitlist control (Active Comparator): An adapted version of the Relaxation Response Resiliency Program (3RP) for parents of children with specific learning disabilities.
  Interventions: Behavioral: Relaxation Response Resiliency Training for Parents of SPLD

INTERVENTIONS:
Behavioral: Relaxation Response Resiliency Training for Parents of SPLD

SUMMARY:
This study has three aims:

Phase I: Through focus group interviews with expert clinicians, leaders of organizations, and parents with children with special needs, this study aims to identify the psychosocial needs of parents of children with learning disabilities, specifically a) the types of concerns that parents find most difficult and stressful b) areas of concern that lack support and resources, and c) areas of need for education and skill training. This study also aims to gather feedback on the Benson-Henry Institute's Relaxation Response Resiliency Program (3RP).

Phase II: Informed by Phase I findings, this study aims to develop and determine the feasibility and acceptability of a virtual 8-session Relaxation Response Resiliency (3RP) program for parents of children with Specific Learning Disabilities (SPLD).

Phase II: This study also aims to test the effectiveness of a pilot wait-list control trial, establishing efficacy of a virtual resiliency program.

DETAILED DESCRIPTION:
According to the 2011/12 National Survey of Children's Health, 14.6 million children in the U.S. have special health care needs (e.g., learning disability, ADD/ADHD, developmental delays, chronic mental or physical health conditions); CSHCN comprise between 14.4%-25.6% of the child population in the United States. Having a child with special health care needs (CSHCN) is associated with an increased risk of problems with emotional and physical health and social well-being. Parents of CSHCN are also at an increased risk for not being employed, financial stress, and poor healthrelated quality of life (HRQoL). There is growing literature on the increased levels of parental stress associated with caring for CSHCN. One study found that chronic stress, as measured by the duration of having a CSHCN, was associated with an increase in clinical aging, determined by telomeres (caps at the end of each strand of DNA that protect chromosomes during aging) sequences. A review article provides a comprehensive overview of the links between high levels of parental stress among parents of children with intellectual and developmental disabilities and child health and well-being. Furthermore, a recent study documented that parents of SSHCN feel socially isolated. Therefore, having a child with special health care needs (CSHCN) is associated with an increased risk of problems with emotional and physical health and social well-being. Parents of CSHCN are also at an increased risk for not being employed, financial stress, and poor health-related quality of life (HRQoL). There is growing literature on the increased levels of parental stress associated with caring for CSHCN, and a recent review article provides a comprehensive overview of the links between high levels of parental stress among parents of children with intellectual and developmental disabilities and child health and well-being.

Resiliency is a multidimensional construct that refers to the ability to maintain adaptation and effective functioning when faced with stressors. Resiliency provides a framework for understanding the adjustment to stress as a dynamic process. Allostasis refers to the capacity to maintain stability of physiological systems in the face of adversity. When the exposed to chronic stressors, such as care for a CSHCN, individuals expend a great deal of energy attempting to maintain allostasis; this can lead to the metabolic wear and tear described as allostatic load. Evidence is accumulating that this wear and tear is mediated by changes in basal stress system activity and by effects of these changes on dependent systems. Allostatic load and resilience can therefore be assessed by measuring basal stress system activity (HPA axis and salivary alpha-amylase). Thus, research to reduce these parents' exposure to stress and, moreover, improve parental responses to stress, may improve the well-being of both parents and their children. Yet, a treatment focused on the psychosocial needs of parents of CSHCN has not been developed. Thus, research is warranted to examine and intervene upon parental stress.

Through focus group interviews with expert clinicians, leaders of organizations, and parents with children with special needs, this study aims to identify the psychosocial needs of parents of children with learning disabilities, specifically a) the types of concerns that parents find most difficult and stressful b) areas of concern that lack support and resources, and c) areas of need for education and skill training. This study also aims to gather feedback on the Benson-Henry Institute's Relaxation Response Resiliency Program (3RP) to advance our next objective to develop a resiliency intervention to provide support to parents of children with learning disabilities. This study aims to evaluate the virtual 3RP for Parents of SPLD in a wait-list control trial and determine a) its feasibility and acceptability and b) its effectiveness at decreasing stress and stress reactivity.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for 3RP intervention:

1. Being the parent of at least one elementary school aged child with a diagnosed specific learning disability
2. Age 18 or older

Exclusion Criteria:

Exclusion criteria for participation in 3RP group:

1. Being the parent of a child with a severe mental or physical disability up to the discretion of the principal investigator
2. Unable or unwilling to sign the informed consent documents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-05-18 (Actual); Study Completion 2018-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elyse Park, PhD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park ER, Perez GK, Millstein RA, Luberto CM, Traeger L, Proszynski J, Chad-Friedman E, Kuhlthau KA. A Virtual Resiliency Intervention Promoting Resiliency for Parents of Children with Learning and Attentional Disabilities: A Randomized Pilot Trial. Matern Child Health J. 2020 Jan;24(1):39-53. doi: 10.1007/s10995-019-02815-3. PMID 31650412

RESULTS

PARTICIPANT FLOW:
Groups:
- 3RP Treatment: An adapted version of the Relaxation Response Resiliency Program (3RP) for parents of children with specific learning disabilities. The adapted program incorporates the three prongs of the 3RP: RR elicitation, stress awareness, and adaptive strategies.
  Relaxation Response Resiliency Training for Parents of SPLD
- Waitlist Control: An adapted version of the Relaxation Response Resiliency Program (3RP) for parents of children with specific learning disabilities.
  Relaxation Response Resiliency Training for Parents of SPLD
Period: Overall Study
Arm/Group | 3RP Treatment | Waitlist Control
Started | 31 | 22
Completed | 19 | 21
Not Completed | 12 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3RP Treatment | Waitlist Control | Total
Number analyzed (Participants) | 31 | 22 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (6.2) | 47 (4.9) | 47 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 48
  Male | 5 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 30 | 21 | 51
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 28 | 20 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Distress
Description: The Visual Analog Scale (VAS)-Distress is a 1-item scale which asks responders to rate their level of distress on a scale of 0 to 10. A higher score indicates more distress.
Time Frame: change between baseline (week 0) to 12 weeks post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3RP Treatment | Waitlist Control
Number analyzed (Participants) | 31 | 22
score on a scale | -1.47 (2.44) | .48 (2.33)

2. Primary Outcome: Current Experiences Scale
Description: The CES is a 25-item measure of resilience adapted from the Post-Traumatic Growth Inventory (PTGI) to reflect current functioning in the domains of appreciation for life (AL), adaptive perspectives (AP), personal strength (PS), spiritual connectedness (SC), relating to others (RO), and an additional four items to assess current adaptive health behaviors (HB) that are not part of the PTGI. The CES is scored on a scale from 0-125 with higher scores indicating greater resilience.
Time Frame: Change between baseline and 12-weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3RP Treatment | Waitlist Control
Number analyzed (Participants) | 31 | 22
score on a scale | 7.67 (7.33) | 1.29 (8.03)

3. Secondary Outcome: Stress Reactivity
Description: The Measure of Current Status Part A (MOCS-A) is a 13-item self-report measure developed to assess participants' current self-perceived status on several skills: the ability to relax at will, recognize stress-inducing situations, restructure maladaptive thoughts, be assertive about needs, and choose appropriate coping responses as needed. Scores can range from 0 to 52, and higher scores are correlated with greater self- perceived proficiency with these skills.
Time Frame: change between baseline (week 0) to 12 weeks post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3RP Treatment | Waitlist Control
Number analyzed (Participants) | 31 | 22
score on a scale | 7.74 (7.59) | -.95 (4.57)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | 3RP Treatment | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/22
Other Adverse Events (participants affected / at risk) | 0/31 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form (2016-09-07): https://cdn.clinicaltrials.gov/large-docs/32/NCT02772432/ICF_000.pdf
  • Study Protocol (2016-09-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT02772432/Prot_001.pdf
  • Statistical Analysis Plan (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/32/NCT02772432/SAP_002.pdf